CLINICAL TRIAL: NCT02579031
Title: A Comparison of an Ultrathin Strut Biodegradable Polymer Sirolimus-Eluting Stent With a Durable Polymer Everolimus-Eluting Stent for Patients With Acute ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Acronym: BIOSTEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 288/15
Record Dates: First submitted 2015-10-16; First posted 2015-10-19 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: Percutaneous Coronary Intervention; Stents; Drug-Eluting Stents; Coronary Artery Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orsiro (Active Comparator): Novel biodegradable-polymer sirolimus-eluting stent Orsiro
  Interventions: Device: Orsiro
- Xience (Active Comparator): Durable-polymer everolimus-eluting stent Xience
  Interventions: Device: Xience

INTERVENTIONS:
Device: Orsiro — Novel biodegradable-polymer sirolimus-eluting stent used during primary percutaneous coronary intervention
  Arms: Orsiro
Device: Xience — Durable-polymer everolimus-eluting stent used during primary percutaneous coronary intervention
  Arms: Xience

SUMMARY:
PCI is considered as the reperfusion strategy of choice for patients with acute STEMI. Data from RCTs and meta-analyses demonstrate a consistent and strong signal towards a significant reduction in MACE among patients with STEMI undergoing primary PCI with newer generation stents with enhanced biocompatibility.

The present trial aims at filling the current gap of evidence by providing randomized data to establish the superior clinical outcome with an ultrathin strut third-generation DES with biodegradable polymer designed to improve vascular healing in patients with STEMI undergoing primary PCI, compared to the current state-of-the art second-generation DES with permanent polymer.

DETAILED DESCRIPTION:
Background

Primary percutaneous coronary intervention (PCI) is considered nowadays as the reperfusion strategy of choice for patients with acute ST-segment elevation myocardial infarction (STEMI, owing to a lower risk of myocardial re-infarction and improved short- and long-term survival compared to fibrinolysis. However, STEMI is still associated with poorer clinical outcomes after PCI, compared to stable CAD, with higher rates of stent thrombosis and an increased risk of myocardial re-infarction persisting throughout long-term follow-up. recent data from randomized controlled trials and meta-analyses demonstrate a consistent and strong signal towards a significant reduction in major adverse cardiac events among patients with STEMI undergoing primary PCI with third-generation DESs, compared with both first-generation and second-generation DESs with durable polymer. Importantly, this signal suggesting superiority of third-generation DESs in patients with STEMI has never been demonstrated with second-generation DESs. Third-generation DESs with enhanced biocompatibility may therefore have a particular clinical benefit in high-risk subgroups of patients with delayed vascular healing but these data warrants confirmation in appropriately designed randomized controlled trials.

Objective

The purpose of the study is to compare the safety and efficacy of a novel biodegradable-polymer sirolimus-eluting stent (Orsiro®) with a durable-polymer everolimus-eluting stent (Xience Xpedition or Xience Alpine®) in a superiority trial among patients presenting with acute STEMI and undergoing primary PCI.

Methods

Eligible patients with acute STEMI presenting within 24 hours of symptom onset will undergo primary PCI. At PCI, the randomly allocated stent has to be implanted in the culprit lesion of the target vessel.

Patients will be followed-up with a hospital visit at 12 months. Patients will be followed-up for clinical endpoints by telephone at 30 days and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ST-segment elevation acute myocardial infarction
* Primary PCI occurring within 24 hours of symptom onset
* Presence of ≥1 acute infarct artery target vessel with one or more coronary artery stenoses in a native coronary artery from 2.25 to 4.0 mm in diameter that can be covered with one or multiple coronary stents

Exclusion Criteria

* Known allergy to aspirin, Ticagrelor, Prasugrel, Clopidogrel, Sirolimus, Everolimus or contrast media
* Planned surgery within 6 months of primary PCI, unless dual antiplatelet therapy could be maintained throughout the peri-surgical period
* Currently participating in another trial before reaching the primary endpoint
* Inability to provide informed consent
* Non-cardiac comorbid conditions with life expectancy of less than 1 year
* Mechanical complication of acute myocardial infarction
* Acute myocardial infarction due to stent thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with target lesion failure (TLF), a composite of cardiac death, target vessel myocardial infarction (Q-wave and non-Q-wave), or clinically driven target lesion revascularization | up to 12 months

SECONDARY OUTCOMES:
Number of patients with clinically indicated and not clinically indicated target lesion revascularization (TLR) | up to 30 days, 1 and 2 years
Number of patients with clinically indicated and not clinically indicated target vessel revascularization (TVR) | up to 30 days, 1 and 2 years
Number of patients with target vessel failure (TVF) | up to 30 days, 1 and 2 years
Number of patients with cardiac death | up to 30 days, 1 and 2 years
Number of patients with all-cause death (cardiac and non-cardiac) | up to 30 days, 1 and 2 years
Number of patients with myocardial infarction (Q-wave and non-Q-wave) | up to 30 days, 1 and 2 years
Number of patients with definite stent thrombosis | up to 30 days, 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, Prof. Dr. med., Principal Investigator — Dep. of Cardiology, Bern University Hospital
Locations (10):
- Switzerland (10):
  - Kantonsspital Aarau, Aarau
  - Universitätsspital Basel, Basel
  - Bern University Hospital, Dep. of Cardiology, Bern
  - Universität Freiburg, Fribourg
  - HUG, Geneva
  - Lausanne University Hospital, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Spital Wallis, Sion
  - Triemli, Zurich

REFERENCES:
- [Result] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Result] Kolh P, Windecker S, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A; European Society of Cardiology Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; EACTS Clinical Guidelines Committee; Sousa Uva M, Achenbach S, Pepper J, Anyanwu A, Badimon L, Bauersachs J, Baumbach A, Beygui F, Bonaros N, De Carlo M, Deaton C, Dobrev D, Dunning J, Eeckhout E, Gielen S, Hasdai D, Kirchhof P, Luckraz H, Mahrholdt H, Montalescot G, Paparella D, Rastan AJ, Sanmartin M, Sergeant P, Silber S, Tamargo J, ten Berg J, Thiele H, van Geuns RJ, Wagner HO, Wassmann S, Wendler O, Zamorano JL; Task Force on Myocardial Revascularization of the European Society of Cardiology and the European Association for Cardio-Thoracic Surgery; European Association of Percutaneous Cardiovascular Interventions. 2014 ESC/EACTS Guidelines on myocardial revascularization: the Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur J Cardiothorac Surg. 2014 Oct;46(4):517-92. doi: 10.1093/ejcts/ezu366. Epub 2014 Aug 29. No abstract available. PMID 25173601
- [Result] Kukreja N, Onuma Y, Garcia-Garcia H, Daemen J, van Domburg R, Serruys PW. Primary percutaneous coronary intervention for acute myocardial infarction: long-term outcome after bare metal and drug-eluting stent implantation. Circ Cardiovasc Interv. 2008 Oct;1(2):103-10. doi: 10.1161/CIRCINTERVENTIONS.108.787762. Epub 2008 Sep 3. PMID 20031664
- [Result] Brodie B, Pokharel Y, Fleishman N, Bensimhon A, Kissling G, Hansen C, Milks S, Cooper M, McAlhany C, Stuckey T. Very late stent thrombosis after primary percutaneous coronary intervention with bare-metal and drug-eluting stents for ST-segment elevation myocardial infarction: a 15-year single-center experience. JACC Cardiovasc Interv. 2011 Jan;4(1):30-8. doi: 10.1016/j.jcin.2010.11.004. PMID 21251626
- [Result] Loh JP, Pendyala LK, Kitabata H, Torguson R, Omar A, Minha S, Chen F, Satler LF, Pichard AD, Waksman R. Comparison of outcomes after percutaneous coronary intervention among different coronary subsets (stable and unstable angina pectoris and ST-segment and non-ST-segment myocardial infarction). Am J Cardiol. 2014 Jun 1;113(11):1794-801. doi: 10.1016/j.amjcard.2014.03.007. Epub 2014 Mar 15. PMID 24837256
- [Result] Nakazawa G, Finn AV, Joner M, Ladich E, Kutys R, Mont EK, Gold HK, Burke AP, Kolodgie FD, Virmani R. Delayed arterial healing and increased late stent thrombosis at culprit sites after drug-eluting stent placement for acute myocardial infarction patients: an autopsy study. Circulation. 2008 Sep 9;118(11):1138-45. doi: 10.1161/CIRCULATIONAHA.107.762047. Epub 2008 Aug 25. PMID 18725485
- [Result] Iqbal J, Sumaya W, Tatman V, Parviz Y, Morton AC, Grech ED, Campbell S, Storey RF, Gunn J. Incidence and predictors of stent thrombosis: a single-centre study of 5,833 consecutive patients undergoing coronary artery stenting. EuroIntervention. 2013 May 20;9(1):62-9. doi: 10.4244/EIJV9I1A10. PMID 23685296
- [Result] Guo N, Maehara A, Mintz GS, He Y, Xu K, Wu X, Lansky AJ, Witzenbichler B, Guagliumi G, Brodie B, Kellett MA Jr, Dressler O, Parise H, Mehran R, Stone GW. Incidence, mechanisms, predictors, and clinical impact of acute and late stent malapposition after primary intervention in patients with acute myocardial infarction: an intravascular ultrasound substudy of the Harmonizing Outcomes with Revascularization and Stents in Acute Myocardial Infarction (HORIZONS-AMI) trial. Circulation. 2010 Sep 14;122(11):1077-84. doi: 10.1161/CIRCULATIONAHA.109.906040. Epub 2010 Aug 30. PMID 20805433
- [Result] Bangalore S, Amoroso N, Fusaro M, Kumar S, Feit F. Outcomes with various drug-eluting or bare metal stents in patients with ST-segment-elevation myocardial infarction: a mixed treatment comparison analysis of trial level data from 34 068 patient-years of follow-up from randomized trials. Circ Cardiovasc Interv. 2013 Aug;6(4):378-90. doi: 10.1161/CIRCINTERVENTIONS.113.000415. Epub 2013 Aug 6. PMID 23922145
- [Result] Otsuka F, Vorpahl M, Nakano M, Foerst J, Newell JB, Sakakura K, Kutys R, Ladich E, Finn AV, Kolodgie FD, Virmani R. Pathology of second-generation everolimus-eluting stents versus first-generation sirolimus- and paclitaxel-eluting stents in humans. Circulation. 2014 Jan 14;129(2):211-23. doi: 10.1161/CIRCULATIONAHA.113.001790. Epub 2013 Oct 25. PMID 24163064
- [Result] Sianos G, Papafaklis MI, Daemen J, Vaina S, van Mieghem CA, van Domburg RT, Michalis LK, Serruys PW. Angiographic stent thrombosis after routine use of drug-eluting stents in ST-segment elevation myocardial infarction: the importance of thrombus burden. J Am Coll Cardiol. 2007 Aug 14;50(7):573-83. doi: 10.1016/j.jacc.2007.04.059. Epub 2007 Jul 30. PMID 17692740
- [Result] Grines CL, Cox DA, Stone GW, Garcia E, Mattos LA, Giambartolomei A, Brodie BR, Madonna O, Eijgelshoven M, Lansky AJ, O'Neill WW, Morice MC. Coronary angioplasty with or without stent implantation for acute myocardial infarction. Stent Primary Angioplasty in Myocardial Infarction Study Group. N Engl J Med. 1999 Dec 23;341(26):1949-56. doi: 10.1056/NEJM199912233412601. PMID 10607811
- [Derived] Haner JD, Rohla M, Losdat S, Iglesias JF, Muller O, Eeckhout E, Kurz D, Weilenmann D, Kaiser C, Tapponnier M, Roffi M, Heg D, Windecker S, Pilgrim T. Ultrathin-strut vs thin-strut drug-eluting stents for multi and single-stent lesions: A lesion-level subgroup analysis of 2 randomized trials. Am Heart J. 2023 Sep;263:73-84. doi: 10.1016/j.ahj.2023.05.004. Epub 2023 May 14. PMID 37192697
- [Derived] Iglesias JF, Muller O, Losdat S, Roffi M, Kurz DJ, Weilenmann D, Kaiser C, Heg D, Windecker S, Pilgrim T. Complex primary percutaneous coronary intervention with ultrathin-strut biodegradable versus thin-strut durable polymer drug-eluting stents in patients with ST-segment elevation myocardial infarction: A subgroup analysis from the BIOSTEMI randomized trial. Catheter Cardiovasc Interv. 2023 Mar;101(4):687-700. doi: 10.1002/ccd.30600. Epub 2023 Feb 19. PMID 36807456
- [Derived] Iglesias JF, Muller O, Losdat S, Roffi M, Kurz DJ, Weilenmann D, Kaiser C, Heg D, Valgimigli M, Windecker S, Pilgrim T. Multivessel percutaneous coronary intervention with thin-strut biodegradable versus durable polymer drug-eluting stents in ST-segment elevation myocardial infarction: A subgroup analysis of the BIOSTEMI randomized trial. Int J Cardiol. 2021 Jul 1;334:37-41. doi: 10.1016/j.ijcard.2021.04.034. Epub 2021 Apr 20. PMID 33887341
- [Derived] Pilgrim T, Muller O, Heg D, Roffi M, Kurz DJ, Moarof I, Weilenmann D, Kaiser C, Tapponnier M, Losdat S, Eeckhout E, Valgimigli M, Juni P, Windecker S, Iglesias JF. Biodegradable- Versus Durable-Polymer Drug-Eluting Stents for STEMI: Final 2-Year Outcomes of the BIOSTEMI Trial. JACC Cardiovasc Interv. 2021 Mar 22;14(6):639-648. doi: 10.1016/j.jcin.2020.12.011. PMID 33727005
- [Derived] Iglesias JF, Muller O, Heg D, Roffi M, Kurz DJ, Moarof I, Weilenmann D, Kaiser C, Tapponnier M, Stortecky S, Losdat S, Eeckhout E, Valgimigli M, Odutayo A, Zwahlen M, Juni P, Windecker S, Pilgrim T. Biodegradable polymer sirolimus-eluting stents versus durable polymer everolimus-eluting stents in patients with ST-segment elevation myocardial infarction (BIOSTEMI): a single-blind, prospective, randomised superiority trial. Lancet. 2019 Oct 5;394(10205):1243-1253. doi: 10.1016/S0140-6736(19)31877-X. Epub 2019 Sep 2. PMID 31488372
- [Derived] Iglesias JF, Roffi M, Degrauwe S, Secco GG, Aminian A, Windecker S, Pilgrim T. Orsiro cobalt-chromium sirolimus-eluting stent: present and future perspectives. Expert Rev Med Devices. 2017 Oct;14(10):773-788. doi: 10.1080/17434440.2017.1378091. Epub 2017 Sep 19. PMID 28889769